CLINICAL TRIAL: NCT02489175
Title: International Prospective Randomized Multicenter Trial to Analyze the Stomaplasty Ring (KoringTM) for Prevention of Parastomal Hernia
Brief Title: Stomaplasty Ring (KoringTM) for Prevention of Parastomal Hernia
Acronym: StoKo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The device used was removed from the market
Sponsor: Nicolas DEMARTINES (Other)
Responsible Party: Sponsor-Investigator, Nicolas DEMARTINES, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202/15
Record Dates: First submitted 2015-06-17; First posted 2015-07-02 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Parastomal Hernia
Keywords: Parastomal hernia; prevention; stomaplasty; ring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stomaplasty KoringTM group (Experimental): The KoringTM is a stomaplasty ring made of propylene, flexible and non-absorbable. It is fixed to the anterior sheath of the abdominal wall in order to prevent PSH.
  Interventions: Device: Stomaplasty KoringTM
- No preventive measure (No Intervention): In these patients, the stoma creation will be traditional, with no mesh implanted

INTERVENTIONS:
Device: Stomaplasty KoringTM — In these patients, the stomaplasty Koring will be implanted at the time of the primary definitive stoma creation. The implantation of the Koring will be performed by experienced surgeons (expertise based, best team approach) who have already implanted the Koring (e.g. participated in the observational study) and/or have reviewed the video documentation. To ensure standardization for all participating centres an operative manual with standardized video sequences is available.
  Arms: Stomaplasty KoringTM group

SUMMARY:
Parastomal hernia (PSH) is one of the most frequent stoma complications with a high impact on patients' quality of life. Half of the stomas created each year are permanent and up to 50% of the patients will develop a PSH. PSH rates depend on the type of ostomy, ileo- or colostomy. End colostomy carries the highest risk for PSH (48%). PSH lead to recurrent pain, poor fitting appliance with leakage and therefore, skin irritation, and can also be complicated by strangulation or occlusion. The literature reports that 30% of patients with a PSH will require surgery. There are many different surgical procedures to repair PSH: primary fascia repair, relocation of the stoma or repair with various type of mesh. Despite the efforts done to improve the techniques, the incidence of recurrent PSH is up to 70% dependent of the used technique. Therefore, the idea of implanting a mesh at the time of initial stoma formation has lately been advocated. A new device, the KoringKM, which is a stomaplasty ring made of propylene, flexible and non-absorbable, was created. This study will try to prove that incorporation of the new stomaplasty ring at the time of stoma creation will diminish long-term PSH rate. This hypothesis will improve patient's quality of life and reduce costs associated with PSH.

All patients requiring a permanent ostomy (ileostomy or colostomy) for a malignant disease and fulfilling the inclusion criteria are eligible to participate in the trial. The patients will be randomized 24 to 48 hours prior to surgery after given written informed consent. The implantation of the Koring will be perfomed by experienced surgeons (expertise based, best team approach) who have already implanted the Koring (e.g. participated in the observational study) and/or have reviewed the video documentation. The surgeon will fill out the first form with the data of the patient and of the surgical procedure. The surgical wound will be daily examined. A second form will be fill out during the 30 post-operative days visit. The patients will be asked to inform the surgeon and/or investigator if any side event or suspicion of infection occurs after hospital discharge. The next follow-up visits will be at one and two years including a clinical examination and an abdominal CT. At this moment, the 3rd and 4th forms will be documented. All data will be anonymised and included in an Excel database.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring permanent ostomy (ileo- or colostomy) for a malignant tumour with at least one year life expectancy
* Patient is able to cooperate
* Patient has given written informed consent
* Age equal or greater than 18 years

Exclusion Criteria:

* Life expectancy < 1 year
* Palliative surgery
* Benign disease
* Factors impacting on the ability to cooperate
* Mental disorders
* Pregnant or breastfeeding women
* Participation in another intervention trial with interference of intervention and outcome of this study
* BMI < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Parastomal hernia rate | at 12 months
  evaluated by abdominal CT and clinical examination, number of patients with parastomal hernia

SECONDARY OUTCOMES:
Stoma necrosis | 30 postoperative days, 12 and 24 months
  Evaluated by clinical examination, number of patients with stoma necrosis
Stoma retraction | 30 postoperative days, 12 and 24 months
  Evaluated by clinical examination, number of patients with stoma retraction
Surgical site infection | 30 postoperative days, 12 and 24 months
  Evaluated by clinical examination, number of patients with surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hahnloser, Professor, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV)
Locations (7):
- Switzerland (7):
  - Cantonal Hospital of Baden, Baden
  - University Hospital of Basel, Basel
  - University Hospital of Geneva, Geneva
  - University Hospital of Lausanne, Lausanne
  - Cantonal Hospital of Schaffhausen, Schaffhausen
  - Limmattal Spital, Schlieren
  - University Hospital of Zürich, Zurich

REFERENCES:
- [Background] Cingi A, Cakir T, Sever A, Aktan AO. Enterostomy site hernias: a clinical and computerized tomographic evaluation. Dis Colon Rectum. 2006 Oct;49(10):1559-63. doi: 10.1007/s10350-006-0681-4. PMID 17120189
- [Background] Londono-Schimmer EE, Leong AP, Phillips RK. Life table analysis of stomal complications following colostomy. Dis Colon Rectum. 1994 Sep;37(9):916-20. doi: 10.1007/BF02052598. PMID 8076492
- [Background] Shabbir J, Chaudhary BN, Dawson R. A systematic review on the use of prophylactic mesh during primary stoma formation to prevent parastomal hernia formation. Colorectal Dis. 2012 Aug;14(8):931-6. doi: 10.1111/j.1463-1318.2011.02835.x. PMID 21929523
- [Background] Cheung MT. Complications of an abdominal stoma: an analysis of 322 stomas. Aust N Z J Surg. 1995 Nov;65(11):808-11. doi: 10.1111/j.1445-2197.1995.tb00566.x. PMID 7487732
- [Background] Hoffmann H, Oertli D, Soysal S, Zingg U, Hahnloser D, Kirchhoff P. A promising new device for the prevention of parastomal hernia. Surg Innov. 2015 Jun;22(3):283-4. doi: 10.1177/1553350614560270. Epub 2014 Nov 27. PMID 25432883
- [Background] Janes A, Cengiz Y, Israelsson LA. Preventing parastomal hernia with a prosthetic mesh: a 5-year follow-up of a randomized study. World J Surg. 2009 Jan;33(1):118-21; discussion 122-3. doi: 10.1007/s00268-008-9785-4. PMID 19011935
- [Background] Hansson BM, Slater NJ, van der Velden AS, Groenewoud HM, Buyne OR, de Hingh IH, Bleichrodt RP. Surgical techniques for parastomal hernia repair: a systematic review of the literature. Ann Surg. 2012 Apr;255(4):685-95. doi: 10.1097/SLA.0b013e31824b44b1. PMID 22418006
- [Background] Janes A, Cengiz Y, Israelsson LA. Experiences with a prophylactic mesh in 93 consecutive ostomies. World J Surg. 2010 Jul;34(7):1637-40. doi: 10.1007/s00268-010-0492-6. PMID 20182719